CLINICAL TRIAL: NCT01767753
Title: A Prospective, Observational, Open Label Study to Assess the 24-hour IOP Fluctuation Pattern Recorded With SENSIMED Triggerfish® in Patients With Primary Open-angle Glaucoma, Before and After Selective Laser Trabeculoplasty
Brief Title: IOP Fluctuations in Patients With Primary Open-angle Glaucoma, Before and After Selective Laser Trabeculoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TF-1207
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Primary Open Angle Glaucoma; Pigmentary Glaucoma; Pseudoexfoliative Glaucoma
Keywords: Glaucoma; SLT
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triggerfish (Experimental): Device: Sensimed Triggerfish
  Interventions: Device: Sensimed Triggerfish

INTERVENTIONS:
Device: Sensimed Triggerfish — Portable investigational device using a contact lens sensor that monitors the IOP fluctuation continuously over 24-hours

SUMMARY:
Selective laser trabeculoplasty (SLT) is an increasingly popular treatment modality in early-to-moderate glaucoma patients. SLT has been suggested to reduce IOP more consistently during the nocturnal period than during the diurnal period in a group of medically-treated patients with primary open angle glaucoma (POAG). At present, there is scarce data on SLT effects on the 24-hour IOP pattern in patients with glaucoma and there is no data on the 24-hour effect of SLT in untreated glaucoma patients.

The purpose of this study is to assess the changes of IOP over a 24-hour period in patients with glaucoma undergoing SLT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open angle glaucoma (POAG) including pigmentary glaucoma or pseudoexfoliative glaucoma (PEX)
* Documented glaucomatous VF damage (in the previous 8 months) with mean defect (MD) > 2.5 dB
* No or stable anti-glaucomatous drug therapy since at least 3 months
* Structural and/or functional glaucomatous damage
* Aged more than 18 years, of either sex
* Not more than 6 diopters spherical equivalent on the study eye
* Not more than 2 diopters cylinder equivalent on the study eye
* Have given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* Refractory glaucoma
* Patients having undergone ocular laser procedures or intraocular surgery for the treatment of glaucoma
* Corneal or conjunctival abnormality precluding contact lens adaptation
* Severe dry eye syndrome
* Patients with allergy to corneal anesthetic
* Patients with contraindications for silicone contact lens wear
* Patients not able to understand the character and individual consequences of the investigation
* Participation in other clinical research within the last 4 weeks
* Any other contra-indication listed in the Triggerfish user manual

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the differences between the nycthemeral IOP patterns recorded with Triggerfish, during two 24-hour periods in patients with POAG, before and after SLT. | 1 months
  * Wake-to-Sleep slopes
  * Overall variability
  * Diurnal and nocturnal IOP patterns
  * Number of peaks

SECONDARY OUTCOMES:
To assess IOP patterns of POAG patients during office hours | 1 month
  Overall variability
  * Diurnal and nocturnal IOP patterns
  * Number of peaks in the study population before and after SLT
Safety and tolerability in this patient population | 1 month
  Adverse events and serious adverse events will be collected throughout the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Nordmann, MD, Principal Investigator — Centre Hospitalier National d'Ophthalmologie des Quinze-Vingts
Locations (1):
- Centre Hospitalier National d'Ophthalmologie des Quinze-Vingts, Paris, France